CLINICAL TRIAL: NCT06114745
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of SHR-1707 in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease and Mild Alzheimer's Disease
Brief Title: A Trial of SHR-1707 Infusion in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease and Mild Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR-1707-103
Record Dates: First submitted 2023-10-11; First posted 2023-11-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer's Disease (AD)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: SHR-1707 injection compared with placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose level 1 SHR-1707 (Experimental): SHR-1707 is administered intravenously.
  Interventions: Drug: SHR-1707 injection
- Dose level 1 Placebo (Placebo Comparator): Placebo is administered intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1707 injection — Drug: SHR-1707 SHR-1707 will be administered through IV infusion. Drug: Placebo Placebo will be administered through IV infusion
  Arms: Dose level 1 SHR-1707
Drug: Placebo — Placebo will be administered through IV infusion
  Arms: Dose level 1 Placebo

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR-1707 in patients with mild cognitive impairment (MCI) due to Alzheimer's disease (AD) and mild AD for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, voluntarily participate in the trial,
2. Male or female aged between 55 years and 85 years (inclusive) at the date of signed consent form.
3. Total body weight of 45~100 kg (inclusive), with a body mass index (BMI) of 19~32 kg/m2 (inclusive)at screening or baseline.
4. The subjects must meet the following clinical criteria for Mild cognitive impairment (MCI) due to Alzheimer's Disease (AD) or criteria for mild AD.
5. The subjects should have a stable caregiver who will help the patients to participate in the whole study process.

Exclusion Criteria:

1. Cognitive impairment due to other medical or neurological factors (non-AD).
2. History of stroke or transient ischemic attack, seizures, or other unexplained loss of consciousness within the past 1 year.
3. Any psychiatric diagnosis that may interfere with the subject's cognitive assessment.
4. Inability to tolerate MRI examination or have contraindications to MRI examination.

6. Exclusion criteria related to previous or concomitant diseases, as listed in the protocol.

7. Exclusion criteria related to general or laboratory tests, as listed in the protocol.

8. The subject is suicidal according to the investigator's judgment or has committed suicidal behaviour within 6 months prior to the screening period.

9. Severe visual or hearing impairment, unable to cooperate in the scale examination.

10. Patients suspected to be allergic to Aβ antibody drugs and their excipients.

11. Women who are pregnant, or women of childbearing age with positive pregnancy test results or are lactating.

12. History of drug abuse and/or drug addiction within 1 year prior to screening.

13 Use of dual antiplatelet or anticoagulant drugs within 3 months prior to the randomization period or planned during the trial.

14.Have had prior treatment with an anti-amyloid immunotherapy within 1 year prior to randomization.

15. Those who have participated in a clinical trial of any drug or medical device within 3 months prior to screening.

16. Investigators and site-related personnel or other persons directly involved in the implementation of the protocol.

17. Other unspecified reasons that, in the opinion of the investigator or sponsor, make the subject unsuitable for enrolment.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Adverse events(AEs) | week 26
  To assess the number of patients with adverse events
Baseline in vital signs value | week 26
  To assess the number of patients with clinically significant change from baseline in vital signs value
Physical examination | week 26
  To assess the number of patients with clinically significant change in physical examination
Laboratory examination | week 26
  To assess the number of patients with clinically significant change from baseline in laboratory examination
Baseline in 12-ECG values | week 26
  To assess the number of patients with clinically significant change from baseline in 12-ECG values
MRI | week 26
  To assess the number of patients with clinically significant change in brain MRI (cerebral edema, microbleeding, etc.)

SECONDARY OUTCOMES:
Aβ positron emission tomography (PET) | week 26
  To assess the change from baseline in intracerebral Aβ deposition as measured by brain Aβ positron emission tomography (PET)
Concentrations of SHR-1707 | week 26
  To assess concentrations of SHR-1707 after multiple doses of administration
Anti-Drug antibody | week 26
  To assess the incidence and time of occurrence of anti-SHR-1707 antibodies

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Liverpool Hospital, Sydney, New South Wales
  - Southern Neurology, Sydney, New South Wales
  - Austin Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No